CLINICAL TRIAL: NCT07008105
Title: Comparing a Single-Session of Cognitive Behavioral Therapy, Pain Reprocessing Therapy, and Emotion Awareness and Expression Therapy for Chronic Pain
Brief Title: Comparing Single-Session Therapies for Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mark A. Lumley (Other)
Responsible Party: Sponsor-Investigator, Mark A. Lumley, Distinguished Professor of Psychology, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-24-10-7277
Record Dates: First submitted 2025-05-14; First posted 2025-06-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic pain; behavioral treatment; CBT; EAET; PRT
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be blinded to condition under after baseline assessment. Outcome assessment will be automated (on-line questionnaires), and thus blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Behavioral Therapy (Experimental): A 90-minute single-session of Cognitive Behavioral Therapy for chronic pain delivered remotely by doctoral students in clinical psychology
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Pain Reprocessing Therapy (Experimental): A 90-minute single-session of Pain Reprocessing Therapy delivered remotely by doctoral students in clinical psychology
  Interventions: Behavioral: Pain Reprocessing Therapy
- Emotion Awareness and Expression Therapy (Experimental): A 90-minute single-session of Emotion Awareness and Expression Therapy delivered remotely by doctoral students in clinical psychology
  Interventions: Behavioral: Emotion Awareness and Expression Therapy
- Treatment As Usual (TAU) (No Intervention): Participants assigned to TAU will not receive any additional psychosocial treatment beyond the other treatments they were receiving before enrolling in this study.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT endorses a pain management model and teaches people skills to cope with chronic pain through reframing thoughts and encouraging behavioral change.
  Arms: Cognitive Behavioral Therapy
Behavioral: Pain Reprocessing Therapy — PRT advocates a pain treatment model in which pain can be substantially reduced by helping people learn that their pain is brain-based and can be substantially reduced or eliminated by decreasing fear of pain and bodily injury and providing education on the neuroscience of pain.
  Arms: Pain Reprocessing Therapy
Behavioral: Emotion Awareness and Expression Therapy — EAET advocates a pain treatment model in which pain can be substantially reduced by helping people learn that their pain is brain-based and can be substantially reduced or eliminated by decreasing fear of pain and of various emotional/interpersonal problems.
  Arms: Emotion Awareness and Expression Therapy

SUMMARY:
Many people in the US suffer from chronic pain. Often times, individuals who have chronic pain also feel depressed, anxious, or hopeless, which can worsen pain. Psychologists, therefore, have developed several treatments to help people with chronic pain. These psychological treatments differ. The most common treatment is Cognitive Behavioral Therapy (CBT) for chronic pain, which helps patients better manage pain through changing thoughts and behaviors. Two newer, less common psychological therapies are Pain Reprocessing Therapy (PRT) and Emotion Awareness and Expression Therapy (EAET). These therapies emphasize that chronic pain is mainly due to plastic processes of over-sensitization in the brain and nervous system, and that psychotherapies can significantly reduce or eliminate pain. Although similar, PRT and EAET stress different aspects of treatment. PRT emphasizes that one's fear of pain and bodily injury maintains the brain's sense of threat, thereby also maintaining the pain response; EAET emphasizes that one's conditioned psychological state of stress and tension maintains a sense of threat, thereby maintaining the pain response. These three treatments have yet to be compared; it is unclear which psychological processes are most important to treating chronic pain.

There is growing interest in single-session psychotherapy interventions. Studies have shown that just a single session of CBT or EAET can help individuals reduce their pain. PRT has yet to be condensed to a single-session intervention.

This study will compare a single session of CBT, PRT, and EAET with a no-treatment control group to test whether 1) one treatment outperforms the others, and 2) different mechanisms/ approaches matter to chronic pain treatment.

DETAILED DESCRIPTION:
Psychological therapies have been found to improve pain and functioning among individuals with chronic pain. Even a single-session of some of these therapies have been found to reduce pain. There are several competing psychological models and therapies for chronic pain that have yet to be compared in a single-session format: Cognitive Behavioral Therapy (CBT), Pain Reprocessing Therapy (PRT), and Emotion Awareness and Expression therapy (EAET). CBT is the most common behavioral intervention for individuals with chronic pain. CBT assists individuals in modulating thoughts and behaviors in order to better manage their pain. However, two newer behavioral treatments for chronic pain, PRT and EAET, postulate that chronic pain can be eliminated, rather than just managed. Both PRT and EAET emphasize that fear underpins pain generation in the nervous system. PRT suggests that fear of injury or further pain maintains chronic pain. EAET suggests that fear of emotional experiences and life stressors maintain chronic pain. These two new therapies, PRT and EAET, have yet to be compared. Individuals with chronic musculoskeletal pain will be randomized to receive either single-session of Cognitive Behavioral Therapy, Pain Reprocessing Therapy, Emotion Awareness and Expression Therapy, or a no-treatment control condition. Participants' pain and mood will be assessed at baseline, pre-intervention, post-intervention, and at two follow-up periods: 1 week and 4 weeks. The purpose of the proposed study is twofold: 1) to compare these three competing models of chronic pain treatment in a single-session, and 2) to investigate what potential mediators of change may be underpinning changes in pain for each treatment. The investigators therefore hypothesize that all 3 treatment types will reduce pain severity and improve functioning; the investigators do not have clear evidence to suggest that one therapy may outperform the others. The secondary hypothesis is that treatment-specific mediators will be more salient in each of the given treatments. The investigators hope to learn what kind of model is most effective for individuals with chronic pain, and whether a single-session of a given intervention can enact meaningful change in pain severity and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Pain for at least 3 months and experienced 4 or more days/week for the past 6 months
* Pain intensity last week is >= 3 (0 to 10 rating scale)
* Pain interference last week is >= 3 (0 to 10 rating scale)
* At least age 18
* Lives in United States
* Fluent in English
* Has personal computer/tablet and internet access
* Able to attend one 90-minute session
* Willing to be randomized
* Seeking to improve their pain-related status via a psychological therapy

Exclusion Criteria:

* Past 2 years (treated for or having experienced):
* Complex regional pain syndrome
* Epilepsy/seizure disorder
* Autoimmune disease
* Liver disease
* Cancer
* Heart disease
* Substance dependence or use disorder
* Schizophrenia or other psychotic disorder
* Bipolar disorder
* Obsessive-compulsive disorder
* Borderline personality disorder
* Suicide attempt or suicide intention or impulse
* Major medical procedure scheduled within next 2 months
* Applied for/ litigating for pain-related disability/worker's compensation (past year).
* Major life event/stressor in past 6 months
* Cognitive impairment (screener score <=4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) - Pain Severity | Baseline to 1-week post-treatment and 1-month follow-up
  4-item measure of pain severity over past week (range 0 to 10; higher scores = worse pain severity)
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference - Short Form 8a | Baseline to 1-week post-treatment and 1-month follow-up
  8-item measure of pain interference over past week (range1 to 5; higher scores = more pain interference)
Pain Rating Question | Immediately pre and immediately post-treatment
  1-item pain rating developed by research team asking "Please rate your pain by circling the one number that tells how much pain you have right now". (0 = No pain, 10 = Pain as bad as you can imagine; higher = more pain)
Symptom Rating Question | Immediately pre and immediately post-treatment
  1 -item symptom rating developed by research team asking "Please rate your physical symptoms by circling the one number that tells how much physical symptoms you have right now". (0 = no symptoms; 10 = symptoms as bad as you can imagine; higher = more symptoms).

SECONDARY OUTCOMES:
Mood Rating Question | Immediately pre and immediately post-treatment
  7-item measure to assess current mood developed by research team asking "For each of the items below, use the 1 to 7 scale and circle a number that indicates how you feel right now". Current mood symptoms assess are: calm, sad, proud, afraid, alert, happy, angry, guilty, nervous on a seven-point scale (1 = not at all, 7 = a great deal; higher = more of that mood)
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function - Short Form 10a | Baseline to 1-week post-treatment and 1-month follow-up
  4-item measure of current physical function (range 1 to 5; higher scores = poorer physical function)
Patient-Reported Outcome Measurement Information System (PROMIS) - Emotional Distress - Anxiety - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  4-item measure of anxiety symptoms in the past week (range 1 to 5; higher scores = more anxiety symptoms)
Patient-Reported Outcome Measurement Information System (PROMIS) - Emotional Distress - Depression - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  4-item measure of depression symptoms in the past week (range 1 to 5; higher scores = more depression symptoms)
Patient Health Questionnaire - Depression | Baseline to 1-week post-treatment and 1-month follow-up
  8-item measure of depression symptoms in the past week (range 0 to 3; higher scores = more depression symptoms)
Patient-Reported Outcome Measurement Information System (PROMIS) - Fatigue - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  4-item measure of fatigue in the past week (range 1 to 5; higher scores = more fatigue)
Patient-Reported Outcome Measurement Information System (PROMIS) - Sleep Disturbance - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  4-item measure of sleep disturbance in the past week (range 1 to 5; higher scores = more sleep disturbance)
Patient-Reported Outcome Measurement Information System (PROMIS) - Emotional Distress - Anger - Short Form 5a | Baseline to 1-week post-treatment and 1-month follow-up
  5-item measure of anger in the past week (range 1 to 5; higher scores = more anger)
Positive and Negative Affect Schedule (PANAS) - Positive Affect - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  5-item measure of positive affect in the past week (range 1 to 5; higher scores = more positive affectivity)
Posttraumatic Stress Disorder Checklist (PCL) - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  5-item measure of trauma symptoms in the past week (range 1 to 4; higher scores = worse PTSD symptoms)
Pain Stages of Change Questionnaire (PSOCQ): Preparation and action | Baseline to 1-week post-treatment and 1-month follow-up
  13-item measure on current readiness to adopt self-management for pain, Preparation and Action items only (range 1 to 5; higher scores = more ready to change)
Opioid Use | Baseline to 1-week post-treatment and 1-month follow-up
  1-item measure on opioid use in past 7 days (range 1 to 7; higher scores = more days)
Employment | Baseline to 1-week post-treatment and 1-month follow-up
  3-item measure on current employment (options for current status and qualitative responses)
Patient Global Impression of Change | 1-week and 1-month follow-up
  1-item measure of overall health change since the start of the study (range 1 to 7; higher scores = more health improvement)
Post-Treatment Satisfaction Questionnaire | 1-week and 1-month follow-up
  8-item measure on patient post-treatment satisfaction (range 1 to 10; higher scores = more satisfied - also included qualitative responses)
Levels of Emotional Awareness Scale (LEAS) - Forms A and B | Baseline to 1-week post-treatment and 1-month follow-up
  10-item measure of current emotional awareness (includes qualitative responses); responses coded for levels of emotional awareness; higher = greater awareness; Form A baseline and Form B at post-treatment
Other Pain Treatments and Health Care Use | Baseline to 1-week post-treatment and 1-month follow-up
  2-item measure of health care currently, the past 6 months, and the past 4 weeks (2 items with yes/no responses and remaining range 0 to 4; higher scores = more treatment)
Inventory of Interpersonal Problems (IIP) | Baseline to 1-week post-treatment and 1-month follow-up
  32-item measure of current interpersonal problems (range 0 to 4; higher scores = more interpersonal problems)
American College of Rheumatology (ACR) Fibromyalgia Diagnostic Criteria - 2011 | Baseline to 1-week post-treatment and 1-month follow-up
  8-item measure on fibromyalgia symptoms in the past week (items with yes/no responses, a checklist, and remaining range 0 to 3; higher scores = worse fibromyalgia symptoms)
Psychological Flexibility Scale (PSYFlex) | Baseline to 1-week post-treatment and 1-month follow-up
  6-item measure of psychological flexibility in the past week (range 0 to 5; higher scores = higher psychological flexibility)
The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool - Part II | Baseline to 1-week post-treatment and 1-month follow-up
  9-item measure on substance use in the past week (yes/no responses); higher scores = more use
Posttraumatic Stress Disorder Checklist (PCL) | Baseline to 1-week post-treatment and 1-month follow-up
  20-item measure of PTSD symptoms (range 0 to 4; higher scores = worse PTSD symptoms)

OTHER OUTCOMES:
Pain Catastrophizing Scale (PCS)-short form | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 6-item measure of pain catastrophizing (range 0 to 4; higher scores = higher pain catastrophizing)
Pain Self-Efficacy Questionnaire (PSEQ) - Short Form | Baseline to 1-week post-treatment and 1-month follow-up.
  Potential Mediator; 4-item measure of current pain self-efficacy (range 0 to 6; higher scores = higher pain self-efficacy)
Survey of Pain Attitudes (SOPA): Pain Control, Disability, Harm, Emotion subscales | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 4, 2-item measures of current pain attitudes (range 0 to 4; higher scores = more of that construct)
Behavioral Activation for Depression (BADS) - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 9-item measure of behavioral activation for depression in the past week (range 0 to 6; higher scores = higher behavioral activation)
Self-Compassion Scale (SCS) - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 12-item measure of situational self-compassion (range 1 to 5; higher scores = less self-compassion)
Chronic Pain Acceptance Questionnaire (CPAQ | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 8-item measure of current chronic pain acceptance (range 0 to 6; higher scores = more chronic pain acceptance)
Chronic Pain Values Inventory (CPVI) | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 6-item measure of current values (checklist responses)
Emotional Approach Coping Scale (EAC) - Short Form | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 4-item measure of emotional approach coping (range 1 to 4; higher scores = higher emotional approach coping)
Emotional Breakthrough Inventory (EBI) | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 6-item measure of emotional breakthroughs in the past week (range 0 to 6; higher scores = more emotional breakthroughs)
Psychological Insight Questionnaire (PIQ) | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 6-item measure of psychological insight in the past week (range 0 to 5; higher scores = more psychological insight)
Brain and Psychological Attributions for Pain | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 9-item measure of current belief of brain and psychological attributions for pain (range 0 to 4; higher scores = higher belief in brain and psychological attributions for pain)
Pain Anxiety Symptom Scale (PASS) | Baseline to 1-week post-treatment and 1-month follow-up
  Potential Mediator; 4-item measure of current pain anxiety symptoms (range 0 to 5; higher scores = worse pain anxiety symptoms)
Adverse Events | Post-treatment and at 1-week and 1-month follow-up
  Potential Mediator; 2-item measure of adverse events in the past week and past month (checklist responses)
Working Alliance Inventory (WAI) - Patient | Immediately post-treatment
  Potential Mediator; 6-item measure of current working alliance (range 0 to 5; higher scores = better working alliance)
Working Alliance Inventory (WAI) - Therapist - Short Form | Immediately post-treatment
  Potential Mediator; 6-item measure of current working alliance (range 0 to 5; higher scores = better working alliance)
Therapist Checklist of Patient Engagement and Homework | Immediately post-treatment
  Potential Mediator; 4-item measure on current patient engagement (range 0 to 8; higher scores = more patient engagement)
Treatment Expectancy and Credibility Questionnaire | Immediately post-treatment
  Potential Mediator; 8-item measure on current treatment expectancy and credibility (range 0 to 10; higher scores = better treatment expectancy)
Evaluation of Therapy Session Rating | Immediately post-treatment
  5-item measure evaluating therapy session and insight (range 1-7; higher scores = higher evaluation)
Manipulation Check | Immediately post-treatment
  9-item measure assessing the degree to which participant's learned intervention-specific material (range 1-7; higher = more information learned)
Demographic / medical history | Baseline
  Potential Moderator: several questions on basic patient background demographics and medical history
Chronic Overlapping Pain Conditions | Baseline
  Potential Moderator: Participants indicate whether they "currently have", "had in the past but not now", or "have never had" a variety of common overlapping pain conditions.
Medication | Baseline
  Potential Moderator: 7-item measure assessing whether patients have taken several different kinds of sleep or pain relief medications within the past 24 hours.
Trauma History Questionnaire - Modified | Baseline
  Potential Moderator: 24-item measure of trauma history, assessing both presence and severity of trauma in childhood and adulthood (range: 0 to 6; higher = more traumatic)
Big Five Inventory, 25-item version | Baseline
  Potential Moderator: 25-items measuring the Big Five personality traits: Neuroticism, Extraversion, Openness, Conscientiousness, Agreeableness (range: 1-5, higher scores = more likely to have a given trait on that subscale)
Multidimensional Scale of Perceived Social Support | Baseline
  Potential Moderator: 12-item measure of perceived social support (range 1 to 7, higher = more support)
Toronto Alexithymia Scale (TAS-20) | Baseline
  Potential Moderator: 20-item measure of alexithymia (range 1 to 5; higher = more alexithymic)
Pain DETECT | Baseline
  Potential Moderator: 7-item screener for neuropathic pain (range: 0 to 5; higher = more likely to have neuropathic pain)
General Pain Treatment Expectancies | Baseline
  Potential Moderator: 3-item measure of expectancy of successful treatment (range 0 to 10, higher = greater expectations)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Wayne State University, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Undecided